CLINICAL TRIAL: NCT03398655
Title: A Randomized, Controlled, Double-Arm, Double-Blind, Multi-Center Study of Ofranergene Obadenovec (VB-111) Combined With Paclitaxel vs. Paclitaxel Combined With Placebo for the Treatment of Recurrent Platinum-Resistant Ovarian Cancer
Brief Title: A Study of VB-111 With Paclitaxel vs Paclitaxel for Treatment of Recurrent Platinum-Resistant Ovarian Cancer (OVAL)
Acronym: OVAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vascular Biogenics Ltd. operating as VBL Therapeutics (Industry)
Collaborators: GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VB-111-701/GOG-3018
Record Dates: First submitted 2018-01-07; First posted 2018-01-12 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2021-06

CONDITIONS: Recurrent Platinum Resistant Ovarian Cancer
Keywords: Recurrent Ovarian cancer; Platinum resistant ovarian cancer; Ovarian cancer; Ovarian carcinoma; Epithelial ovarian cancer; paclitaxel
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): VB-111 + Paclitaxel
  Interventions: Drug: VB-111 + Paclitaxel
- Arm 2 (Active Comparator): Placebo + Paclitaxel
  Interventions: Drug: Placebo + Paclitaxel

INTERVENTIONS:
Drug: VB-111 + Paclitaxel — VB-111 will be administered intravenously at a dose of 1x10e13 VPs every 2 months Paclitaxel will be administered intravenously at a dose of 80mg/m2 every week
  Other Names: Ofranergene Obadenovec
  Arms: Arm 1
Drug: Placebo + Paclitaxel — Placebo will be administered intravenously every 2 months Paclitaxel will be administered intravenously at a dose of 80mg/m2 every week
  Arms: Arm 2

SUMMARY:
The purpose of this phase 3, randomized, multicenter study is to compare VB-111 and paclitaxel to placebo and paclitaxel in adult patients with Recurrent Platinum-Resistant Ovarian Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients ≥18 years of age
2. Histologically confirmed epithelial ovarian cancer and documented disease.
3. Patients must have platinum-resistant disease
4. Patients must have disease that is measurable according to RECIST 1.1 and require chemotherapy treatment.
5. ECOG PS 0-1.
6. Adequate hematological functions:

   * ANC ≥ 1000/mm3
   * PLT ≥ 100,000/mm3
   * PT and PTT (seconds) < 1.2 X ULN. Patients who are anticoagulated do not need to meet criteria for PT and PTT.
7. Patients who are known to carry a BRCA mutation may be enrolled only after (following PARP inhibitor treatment failure, or being intolerant of, or ineligible for PARP inhibitor treatment).

Exclusion Criteria:

1. Non-epithelial tumors (Carcino-sarcomas are excluded)
2. Ovarian tumors with low malignant potential (i.e. borderline tumors) clear cell carcinomas, grade 1 serous tumors or mucinous tumors.
3. History of other clinically active malignancy within 5 years of enrollment, except for tumors with a negligible risk for metastasis or death, such as adequately controlled basal-cell carcinoma, adequately controlled, non-metastatic squamous-cell carcinoma of the skin, or carcinoma in situ of the cervix or breast.
4. Previous ovarian cancer treatment with >5 anticancer regimens.
5. Any prior radiotherapy to the pelvis or whole abdomen.
6. Inadequate liver function, defined as serum creatinine > ULN, unless calculated creatinine clearance > 50ml/min (by Cockroft & Gault formula):

   * Serum (total) bilirubin > ULN (Exception: documented Gilbert's disease patients can be enrolled)
   * Alkaline phosphatase, AST/SGOT or ALT/SGPT ≥2.5 x ULN (or ≥ 5 x ULN in the presence of liver metastases).
7. Inadequate renal function, defined as:

   * Serum creatinine > ULN OR
   * Calculated creatinine clearance < 50ml/min (by Cockroft & Gault formula)
8. New York Heart Association (NYHA) Grade II or greater congestive heart failure
9. History of myocardial infarction or unstable angina within 6 months prior to day of randomization.
10. History of stroke or transient ischemic attack within 6 months prior to day of randomization.
11. Patient with proliferative and/or vascular retinopathy
12. Known brain metastases
13. History of hemoptysis or active GI bleeding within 6 month prior to day of randomization
14. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
15. History of abdominal fistula or gastrointestinal perforation.
16. Current signs and symptoms of bowel obstruction
17. Uncontrolled active infection
18. Patients who had evidence of disease progression during or up to 90 days from the last dose of the first line of platinum based therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 408 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Overall Survival | From randomization until death from any cause (up to 5 years after last study treatment)
Progression Free Survival (PFS) by RECIST 1.1 | From randomization until progression defined according to RECIST 1.1 or death, whichever occurs first (up to 5 years after last study treatment)

SECONDARY OUTCOMES:
Combined CA-125 and RECIST 1.1 response (GCIG) | From date of study entry until the date of death from any cause, or up to 5 years after last study treatment
CA-125 Response (GCIG) | From date of study entry until the date of death from any cause, or up to 5 years after last study treatment
Objective response rate (ORR) by RECIST 1.1 | From date of study entry until the date of death from any cause, or up to 5 years after last study treatment
OS100 for a sensitivity analysis of OS | From 100 days after date of study entry until the date of death from any cause, or up to 5 years after last study treatment

CONTACTS AND LOCATIONS:
Locations (94):
- United States (64):
  - UAB Division of GYN Oncology, Birmingham, Alabama
  - Western Regional Medical Center, Goodyear, Arizona
  - Arizona Oncology Associates, PC - HAL - USO, Phoenix, Arizona
  - Arizona Oncology Associates, PC - HAL - USO, Tempe, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - UCLA-JCCC-Women's Health Clinical Research Unit, Los Angeles, California
  - The Center for Cancer Prevention and Treatment at St. Joseph Hospital of Orange, Orange, California
  - University of California, Irvine Medical Center/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California - San Francisco, San Francisco, California
  - Sansum Clinic - USO, Santa Barbara, California
  - Olive View UCLA Medical Center, Sylmar, California
  - Hartford HealthCare Cancer Institute at the Hospital of Central Ct, Hartford, Connecticut
  - Hartford Healthcare, Hartford, Connecticut
  - UF Health, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Midwestern Regional Medical Center, Inc, Zion, Illinois
  - Parkview Cancer Institute, Fort Wayne, Indiana
  - Indiana University School of Medicine, Indianapolis, Indiana
  - St. Vincent Gynecologic Oncology, Indianapolis, Indiana
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Hospital, Detroit, Michigan
  - Dartmouth- Hitchcock Medical Center, Lebanon, New Hampshire
  - Atlantic Health System/Morristown Medical Center, Morristown, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Women's Cancer Care Associates, LLC, Albany, New York
  - Westchester Medical Center, Hawthorne, New York
  - Northwell Health Cancer Institute, Lake Success, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Health Quest Medical Practice, Division of Gynecology/Oncology Gyno Dyson Cancer Center Vassar Brothers Medical Center, Poughkeepsie, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Duke University-Duke Cancer Institute, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Sanford Medical Center, Fargo, North Dakota
  - University of Cincinnati, Cincinnati, Ohio
  - Womens Cancer Center/Kettering Cancer Care, Kettering, Ohio
  - University of Oklahoma Health Sciences Center-Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - The University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - GHS Cancer Institute, Greenville, South Carolina
  - Sanford Clinical Research, Sioux Falls, South Dakota
  - Texas Oncology, Austin Central - USO, Austin, Texas
  - Memorial Hermann, Houston, Texas
  - UT Health, San Antonio, Texas
  - Universtiy of Vermont, Burlington, Vermont
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Marshfield Clinic Cancer Care & Research Center, Marshfield, Wisconsin
  - Froedtert and Medical College of Wisconsin, Milwaukee, Wisconsin
- Israel (6):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Shaare Tzedek Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Department of Oncology, Rehovot
- Japan (12):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Ehime University Hospital, Tōon, Ehime
  - Kurume University Hospital, Kurume, Fukuoka
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Iwate Medical University Hospital, Shiwa-gun, Iwate
  - Tohoku University Hospital, Sendai, Myagi
  - National Defense Medical College Hospital, Tokorozawa, Saitama
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto, Tokyo
  - Niigata Cancer Center Hospital, Niigata
  - Hokkaido University Hospital, Sapporo
- Poland (3):
  - Centrum Badan Klinicznych Jagiellonskiego Centrum Innowacji, Krakow
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej MSWiA z Warminsko-Mazurskim Centrum Onkologii w Olsztynie, Olsztyn
  - MedPolonia Sp. z o.o., Poznan
- Spain (9):
  - Parc Taulí Hospital Universitari Edifici Santa Fe, Planta 0, Sala de recerca 3, Barcelona
  - Institut Català d'Oncologia - Hospital Duran i Reynals, Barcelona
  - Hospital Universitario de Donostia Edificio Onkologikoa- Planta baja, Sala de Ensayos Clinicos, Donostia / San Sebastian
  - Hospital Gregorio Marañon Módulo prefabricado Oncología, Planta Baja, Madrid
  - MD Anderson Cancer Center Madrid Unidad de ensayos Clinicos, Madrid
  - Hospital Universitario Clínico San Carlos., Madrid
  - Hospital Universitario Virgen del Rocío Servicio Oncología Médica. Ensayos Clínicos. Edificio CDCA, Seville
  - Instituto Valenciano de Oncología Médica (IVO, Valencia
  - Consorcio Hospitalario General Universitario de Valencia Servicio de Oncología Médica - Unidad de Investigación, Valencia

REFERENCES:
- [Derived] Arend RC, Monk BJ, Shapira-Frommer R, Haggerty AF, Alvarez EA, Amit A, Alvarez Secord A, Muller C, Casado Herraez A, Herzog TJ, Tewari KS, Cohen JG, Huang M, Yachnin A, Holeman LL, Ledermann JA, Rachmilewitz Minei T, Buyse M, Fain Shmueli S, Lavi M, Harats D, Penson RT; OVAL/GOG-3018 Investigators. Ofranergene Obadenovec (Ofra-Vec, VB-111) With Weekly Paclitaxel for Platinum-Resistant Ovarian Cancer: Randomized Controlled Phase III Trial (OVAL Study/GOG 3018). J Clin Oncol. 2024 Jan 10;42(2):170-179. doi: 10.1200/JCO.22.02915. Epub 2023 Oct 31. PMID 37906726
- [Derived] Arend RC, Monk BJ, Herzog TJ, Moore KN, Shapira-Frommer R, Ledermann JA, Tewari KS, Secord AA, Rachmilewitz Minei T, Freedman LS, Miller A, Shmueli SF, Lavi M, Penson RT. Utilizing an interim futility analysis of the OVAL study (VB-111-701/GOG 3018) for potential reduction of risk: A phase III, double blind, randomized controlled trial of ofranergene obadenovec (VB-111) and weekly paclitaxel in patients with platinum resistant ovarian cancer. Gynecol Oncol. 2021 May;161(2):496-501. doi: 10.1016/j.ygyno.2021.02.014. Epub 2021 Feb 23. PMID 33637348
- See also: VBL Therapeutics Company Website — http://www.vblrx.com/